CLINICAL TRIAL: NCT05373524
Title: Rheopheresis Mechanism of Action and Impacts on the Evolution of Peripheral Arterial Disease in Hemodialysis Patients
Brief Title: Rheopheresis Mechanism in Hemodialysis Patients With PAD
Acronym: VALLOIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC20.461
Record Dates: First submitted 2022-01-18; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Intervention Model Description: Rheopheresis procedure/Shamapheresis procedure
Who Masked: Investigator
Masking Description: The efficacy will be assessed by a vascular surgeon blinded to the study group during consultation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the rheopheresis group (Active Comparator): Rheopheresis is performed using an automated monitor in a double-filtration cascade. Plasma purify from of high molecular weight proteins through a secondary filter is then returned to the patient. This technique is performed in tandem with a hemodialysis monitor.
  Interventions: Biological: Biological analysis
- the shamapheresis group (Placebo Comparator): Shamapheresis is performed with the same automated monitor (Plasauto, HemaT company). Extracted plasma is not treated through the secondary filter (Rheofilter) and return to the patient. This technique is performed in tandem with a hemodialysis monitor.
  Interventions: Biological: Biological analysis

INTERVENTIONS:
Biological: Biological analysis — Rheopheresis using plasma separation and plasma filtration, coupled to hemodialysis

SUMMARY:
Peripheral arterial disease (PAD) is common in chronic hemodialysis patients (HDC) with a prevalence of 30% according to the DOPPS study.

The combination of PAD and chronic kidney disease (CKD) stage 5 is a risk factor for major amputation (24.5%) with a mortality rate of 55% at 2 years.

Ischemia occurring during PAD is the result of impaired microcirculation, with insufficient blood flow to maintain tissue perfusion and viability.

It is responsible for painful skin wounds whose healing is poor, with a significant risk of infection.

In patients with chronic renal failure, it is linked to both:

* local phenomena (atherosclerosis, calcification)
* changes in blood viscosity (elevated hematocrit and inflammatory proteins, especially fibrinogen)
* a neovascularization defect (uremic toxins, in particular indoxyl sulphate). If revascularization is not possible, amputation remains the only possible treatment to relieve pain and limit the risk of infection.

Rheopheresis is an apheresis technique that allows the depletion of high molecular weight serum proteins.

This would reduce blood viscosity and red blood cell (RBC) aggregation, thereby improving microvascular perfusion, with the aim of reducing pain, improving healing and limiting the risk of amputation.

Several studies have investigated the efficacy of rheopheresis in PAD in HDC, but the level of evidence remains low.

DETAILED DESCRIPTION:
The main objective of our study is to evaluate the impact of rheopheresis on blood (main objective) and plasma viscosity, skin microcirculation and blood coagulation (Fibrinography, Thrombin Generation).

No study has evaluated the direct effect of rheopheresis on these different parameters.

However, a better understanding of these mechanisms would make it possible both to optimize the effectiveness of the technique, to limit its potential side effects and the cost of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more and included in the RHEOPAD protocol (2019-A01513-54)
* ESRD treated by hemodialysis or hemodiafiltration
* PAD-LTI with tissue loss and/or wounds (ulcers or gangrene) with at least one of the following criterion, subject to the feasibility of the measures: arterial pressure assessment at the ankle <70 mmHg, or toe pressure 30 mm Hg, or transcutaneous oximetry measurements < 40 mm Hg
* Interventional or surgical revascularization either not technically possible or no necessary
* Medical insurance
* Signed informed consent

Exclusion Criteria:

* - Uncontrolled infection despite well-conducted antibiotic therapy
* Life expectancy < 1 year
* Severe cognitive or psychiatric disorders
* Pregnant woman, parturient, nursing mother
* Patients unable to give an informed consent or unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in Blood viscosity measured by rotational rheometer | Immediately before 1ST and immediately after 12th procedure , outcome measurement will be reported at the end of the study (approximately 3 years)
  To assess the effect of rheopheresis on blood viscosity of chronic hemodialysis patients with PAD

SECONDARY OUTCOMES:
Blood viscosity measured by rotational rheometer | up to 24 weeks
  Evaluate the effect of rheopheresis on blood viscosity measured by rotational rheometer before the 12th treatment session

OTHER OUTCOMES:
Evaluate the effect of rheopheresis on plasma viscosity measured by falling ball viscometer | Immediately before day 0 and 12-th procedure and immediately after 1st procedure
  Plasma viscosity measured by falling ball viscometer in pre vs post session 1 and in pre session 12 vs baseline.
Evaluate the effect of rheopheresis on skin microvascular function (1st and 12th sessions pre and post session) | Immediately before day0 and 1 years
  Post-occlusive and thermal hyperaemia of cutaneous blood flow measured by speckle contrast imaging, compared between the rheopheresis and shamapheresis groups (1st and 12th sessions pre and post session)
Evaluate the effect of rheopheresis on coagulation | Immediately before day 0 and 12-th procedure and immediately after 1st procedure
  Study of the lifespan of the blood clot (difference between formation time and clot lysis time) using a multi-well plate spectrophotometer (Fibrinography);

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roustit M, Cracowski JL. Assessment of endothelial and neurovascular function in human skin microcirculation. Trends Pharmacol Sci. 2013 Jul;34(7):373-84. doi: 10.1016/j.tips.2013.05.007. Epub 2013 Jun 21. PMID 23791036
- [Result] Meyer A, Fiessler C, Stavroulakis K, Torsello G, Bisdas T, Lang W; CRITISCH collaborators. Outcomes of dialysis patients with critical limb ischemia after revascularization compared with patients with normal renal function. J Vasc Surg. 2018 Sep;68(3):822-829.e1. doi: 10.1016/j.jvs.2017.12.048. Epub 2018 Mar 26. PMID 29598891
- [Result] Lowry D, Saeed M, Narendran P, Tiwari A. The Difference Between the Healing and the Nonhealing Diabetic Foot Ulcer: A Review of the Role of the Microcirculation. J Diabetes Sci Technol. 2017 Sep;11(5):914-923. doi: 10.1177/1932296816658054. Epub 2016 Jul 10. PMID 27390224
- [Result] Weiss N. A critical review on the use of lipid apheresis and rheopheresis for treatment of peripheral arterial disease and the diabetic foot syndrome. Semin Dial. 2012 Mar-Apr;25(2):220-7. doi: 10.1111/j.1525-139X.2011.01036.x. Epub 2011 Dec 16. PMID 22175277
- [Result] Ferrannini M, Vischini G, Staffolani E, Scaccia F, Miani N, Parravano MC, Louis MM, Splendiani G, Di Daniele N. Rheopheresis in vascular diseases. Int J Artif Organs. 2007 Oct;30(10):923-9. doi: 10.1177/039139880703001010. PMID 17992654
- [Result] Klingel R, Mumme C, Fassbender T, Himmelsbach F, Altes U, Lotz J, Pohlmann T, Beyer J, Kustner E. Rheopheresis in patients with ischemic diabetic foot syndrome: results of an open label prospective pilot trial. Ther Apher Dial. 2003 Aug;7(4):444-55. doi: 10.1046/j.1526-0968.2003.00082.x. PMID 12887730
- [Result] Kirschkamp T, Schmid-Schonbein H, Weinberger A, Smeets R. Effects of fibrinogen and alpha2-macroglobulin and their apheretic elimination on general blood rheology and rheological characteristics of red blood cell aggregates. Ther Apher Dial. 2008 Oct;12(5):360-7. doi: 10.1111/j.1744-9987.2008.00610.x. PMID 18937718
- [Result] Briers JD. Laser Doppler, speckle and related techniques for blood perfusion mapping and imaging. Physiol Meas. 2001 Nov;22(4):R35-66. doi: 10.1088/0967-3334/22/4/201. PMID 11761081
- [Result] Roustit M, Millet C, Blaise S, Dufournet B, Cracowski JL. Excellent reproducibility of laser speckle contrast imaging to assess skin microvascular reactivity. Microvasc Res. 2010 Dec;80(3):505-11. doi: 10.1016/j.mvr.2010.05.012. Epub 2010 Jun 9. PMID 20542492
- [Result] Choi B, Ramirez-San-Juan JC, Lotfi J, Stuart Nelson J. Linear response range characterization and in vivo application of laser speckle imaging of blood flow dynamics. J Biomed Opt. 2006 Jul-Aug;11(4):041129. doi: 10.1117/1.2341196. PMID 16965157
- [Result] Stewart CJ, Frank R, Forrester KR, Tulip J, Lindsay R, Bray RC. A comparison of two laser-based methods for determination of burn scar perfusion: laser Doppler versus laser speckle imaging. Burns. 2005 Sep;31(6):744-52. doi: 10.1016/j.burns.2005.04.004. PMID 16129229